CLINICAL TRIAL: NCT04888871
Title: Randomized Control Trial for Comparison of Prevention and Appropiate Obstetric Interventions for Prolonged Second Stage Labor at Term Pregnancies During Vaginal Delivery
Brief Title: Comparison of Prevention and Appropiate Obstetric Interventions for Prolonged Second Stage Labor at Term Pregnancies During Vaginal Delivery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Resul Karakuş, Specialist, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Other Study IDs: 2020/123
Record Dates: First submitted 2021-05-11; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Obstetric Labor Complications; Vacuum Extraction; Failure, Affecting Fetus or Newborn; Complicated Labour/Delivery Livebirth
Keywords: labor stage, second
MeSH Terms: conditions — Obstetric Labor Complications; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Only Fundal Pressure (Kristeller Maneuver): prolonged second stage phase and not prolonged second phase in pregnant women to singletons at the weeks between 37-42, applying Only Fundal Pressure (Kristeller Maneuver) and the postpartum evaluation of maternal episiotomy needs presence of second and third degree perineal tears, presence of postpartum hemorrhage and need for blood transfusion , cesarean rates and fetal first and fifth minute Apgar score , fetal blood gas parameters, presence of fetal trauma, need for neonatal intensive care will
- Only Vacuum Extraction: prolonged second stage phase and not prolonged second phase in pregnant women to singletons at the weeks between 37-42, applying only vacuum extraction and the postpartum evaluation of maternal episiotomy needs presence of second and third degree perineal tears, presence of postpartum hemorrhage and need for blood transfusion , cesarean rates and fetal first and fifth minute Apgar score , fetal blood gas parameters, presence of fetal trauma, need for neonatal intensive care will
- Both Fundal Pressure (Kristeller Maneuver) and Vacuum Extraction: prolonged second stage phase and not prolonged second phase in pregnant women to singletons at the weeks between 37-42, applying Both Fundal Pressure (Kristeller Maneuver) and Vacuum Extraction and the postpartum evaluation of maternal episiotomy needs presence of second and third degree perineal tears, presence of postpartum hemorrhage and need for blood transfusion , cesarean rates and fetal first and fifth minute Apgar score , fetal blood gas parameters, presence of fetal trauma, need for neonatal intensive care will

SUMMARY:
Randomized Control Trial for Comparison of Prevention and Appropiate Obstetric Interventions for Prolonged Second Stage Labor at Term Pregnancies During Vaginal Delivery.

DETAILED DESCRIPTION:
This study includes prolonged second stage phase and not prolonged second phase in pregnant women to singletons at the weeks between 37-42. Fetal head level will be at or below the ischial spines in all patients.Patients with fully dilated cervix will be included in the study and the bladder will be emptied completely on the labor table. Patients diagnosed with fetal distress will not be included in the study.Indicated patients will be randomly divided into three groups; one group will be only subjected to a Fundal Pressure (Kristaller Maneuver), second group will only be subjected to Vacuum Extraction and the third group will be subjected to both Fundal Pressure (Kristaller Maneuver) and Vacuum Extraction. Maternal episiotomy needs presence of second and third degree perineal tears, presence of postpartum hemorrhage and need for blood transfusion , cesarean rates and fetal first and fifth minute Apgar score , fetal blood gas parameters, presence of fetal trauma, need for neonatal intensive care will be evaluated among three randomized groups.

ELIGIBILITY:
Inclusion Criteria:

* term pregnancy weeks between 37-42, singleton, vertex presentations
* prolonged second stage of labor
* Fetal head is minimum at the level of ischial spin
* maternal incompatibility during/after second stage of labor
* complete cervical dilatation

Exclusion Criteria:

* Fetal distress
* Uncomplete cervical dilatation
* twin pregnancies or polycyesia
* Pregnancy weeks lower than 37weeks
* other than vertex presentations
* Fetal Anomalies

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Study Population: Randomized Control Trial for Comparison of Prevention and Appropiate Obstetric Interventions for Prolonged Second Stage Labor at Term Pregnancies During Vaginal Delivery.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
maternal morbidity | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Kamil Maternity and Childrens Hospital, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No